CLINICAL TRIAL: NCT06210308
Title: Preoperative Ultrasound Evaluation of Gastric Contents in Voluntary Termination of Pregnancy (IVG) During the First Trimester: Prospective Observational Study of Patients With Gestational Nausea and Vomiting
Brief Title: Preoperative Ultrasound Evaluation of Gastric Contents in Voluntary Termination of Pregnancy During the First Trimester
Acronym: ECHONAV
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-13Obs-CHRMT
Record Dates: First submitted 2024-01-04; First posted 2024-01-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Voluntary Termination of Pregnancy
Keywords: Voluntary Termination of Pregnancy; Preoperative gastric content

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Data collection from gastric ultrasound — observational study

SUMMARY:
This is an observational, prospective, monocentric, diagnostic study aiming to evaluate the diagnostic properties of the presence of nausea-vomiting in predicting the existence of gastric contents in preoperative surgical abortion.

DETAILED DESCRIPTION:
Most surgical abortions are performed under general anaesthesia. Inhalation of gastric contents is one of the main complications of general anesthesia, in terms of frequency and severity. Patients in the 1st trimester of pregnancy are frequently subject to nausea and vomiting, even on an empty stomach. The presence of nausea and vomiting prior to surgery means that the anesthetic protocol needs to be modified, as there is a greater risk of complications, particularly allergic ones. Preoperative gastric ultrasound is recognized for its ability to predict the risk of gastric inhalation during anesthesia. It is a non-irradiating, non-invasive, painless and rapid examination. There are no data on the association between gestational nausea and vomiting and the risk of inhalation in the context of preoperative fasting. There are no data on the gastric volume of patients in the 1st trimester of pregnancy with or without nausea. Does gestational nausea and vomiting represent an anesthetic risk of gastric inhalation?

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Patients undergoing Voluntary termination of pregnancy by dilatation and aspiration before 14 weeks of amenorrhea

Exclusion Criteria:

* Patient under guardianship or curatorship.
* Patient with language barrier.
* Any condition causing the patient to be considered as having a "full stomach" even before the gastric ultrasound:

  * body mass index (BMI) > 40 kg/m2
  * Hiatal hernia.
  * History of gastric or esophageal surgery or neoplasia.
  * Gastroparesis (diabetic, hepatocellular insufficiency, severe renal insufficiency, etc.).
* Opposition of the patient to the re-use of her data for the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Voluntary termination of pregnancy by dilatation and aspiration before 14 weeks of amenorrhea
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Prediction of gastric content by ultrasound | Day 0
  according to the presence of nausea or vomiting : Sensitivity, specificity, positive and negative predictive values

SECONDARY OUTCOMES:
Prevalence of presence of gastric content | Day 0
  Solid / liquid / none
nausea or vomiting | Day 0
  Presence of nausea or vomiting on the day of surgery, or use of anti-nausea medication during pregnancy
Anesthesia protocol | Day 0
  incidence of modification of anesthesia protocol consecutive of the realization of gastric ultrasound
Respiratory complications | At discharge from the recovery room up to one hour
  any respiratory complications that may have occurred during the operation, right up to the time of discharge from the recovery room

CONTACTS AND LOCATIONS:
Overall Officials: Léo COINUS, MD, Principal Investigator — CHR Metz Thionville Hopital Mercy
Locations (1):
- CHR Metz-Thionville/Hopital Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No
According to the French law and the French Data Protection Authority (CNIL), we won't be able to publicly share individual participant data, but we plan to share their conclusions through peer-reviewed publications and conferences.